CLINICAL TRIAL: NCT05172999
Title: A Randomized Controlled Pilot Study of Polyethylene Glycol Loxenatide Plus LNG-IUS in Women With Endometrial Atypical Hyperplasia
Brief Title: Loxenatide Plus LNG-IUS in Endometrial Atypical Hyperplasia
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaojun Chen, Principal Investigator，Clinical Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53211033
Record Dates: First submitted 2021-12-12; First posted 2021-12-29 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Atypical Endometrial Hyperplasia; Obesity; Fertility Issues
Keywords: atypical endometrial hyperplasia, obesity, fertility
MeSH Terms: conditions — Endometrial Hyperplasia; Obesity; Infertility | interventions — polyethylene glycol loxenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LNG-IUS (Active Comparator): enrolled patients will receive LNG-IUS for 6 months or longer till complete response
  Interventions: Device: levonorgestrel-releasing intrauterine system
- LOX+LNG-IUS (Experimental): enrolled patients will receive LNG-IUS plus polyethylene glycol loxenatide for treatment.
  Interventions: Device: levonorgestrel-releasing intrauterine system; Drug: Polyethylene Glycol Loxenatide

INTERVENTIONS:
Device: levonorgestrel-releasing intrauterine system — Enrolled patients will be inserted this device for treating AEH to preserve fertility for 3-6 months or longer till complete response or operation if treatment fails, and the device may be removed if treatment changes.
  Other Names: MIRENA
Drug: Polyethylene Glycol Loxenatide — Initiate injection of Loxenatide will be 0.1mg per week, if the patient can tolerate, the dose will be increased to 0.2mg per week, or else 0.1mg per week will be injected and the injection will last for no more than 28 weeks. If the patient cannot tolerate the least 0.1mg/week, she must be excluded from this trial.
  Other Names: Fulaimei; PEX168
  Arms: LOX+LNG-IUS

SUMMARY:
To study if polyethylene glycol loxenatide plus levonorgestrel-releasing intrauterine system (LNG-IUS) will improve response rates in patients with endometrial atypical hyperplasia.

DETAILED DESCRIPTION:
Background: Obesity or overweight is associated with lower treatment response and longer time to achieve complete response(CR) in patients with atypical endometrial hyperplasia (AEH) who want to preserve fertility, as evidenced by our research and lots of published studies. The larger the baseline weight of AEH patients, the more the weight gains after high-dose progesterone treatment. Obese AEH patients have a lower response to high-dose progesterone.

Losing weight may help improve treatment response. Weight management and lifestyle intervention have been written into 2020 uterine NCCN (National Comprehensive Cancer Network) guidelines. Our research showed that metformin may improve insulin resistance in patients with AEH, and shorten time to achieve CR, and increase the CR rates. Theoretically, Losing weight can improve the chronic inflammatory environment in the endometrium and whole body and improve metabolic disorder which help patients achieve CR.

LNG-IUS will be adopted in this research. Though LNG-IUS and high-dose progesterone have similar efficacy in treating AEH patients, long-term treatment of progesterone has many side effects. Compared to oral progesterone, LNG-IUS has fewer side effects and fewer effects on weight gaining.

GLP-1 receptor agonist (GLP-1RA), which is one of the commonly used hypoglycemic drugs, has been approved for weight control. Loxenatide is the first Chinese-produced long-acting GLP-1R agonist. It is applicable for diabetes patients. In the USA, some GLP-1RA has been applied for losing weight, such as liraglutide and semaglutide. GLP-1RA acts through improving insulin sensitivity, decreasing glucagon secretion, inhibiting appetite, delaying gastric emptying, and improving whole-body inflammation condition. Loxenatide plus LNG-IUS may improve the efficacy of preserving fertility in obese AEH patients through help patients lose weight.

Objective: To investigate whether loxenatide plus LNG-IUS improves the efficacy of preserving fertility when compared to LNG-IUS alone in obese women with AEH who want fertility conservation.

Design: A pilot prospective randomized controlled study is designed. And this study is open-label. We use SPSS software (version 22.0, IBM) to perform simple randomization and get randomized numbers. And participants will be randomly assigned (1:1) to receive LNG-IUS alone or loxenatide plus LNG-IUS. Patients in LNG-IUS alone group will accept LNG-IUS insertion as treatment and the other group cases will be treated with loxneatide plus LNG-IUS.

All enrolled patients will receive basic medical treatment in weight management and lifestyle improvement support, no enhanced interventions. Hysteroscopic assessment, metabolic and inflammatory indications will be performed every 12-16 weeks, while other indexes (weight, body composition change, side effects, and so on) will be evaluated every month.

For the efficacy evaluation, CR is defined as the reversion of endometrial atypical hyperplasia to proliferative or secretory endometrium; partial response (PR) is defined as regression to simple or complex hyperplasia without atypia; no response (NR) is defined as the persistence of the disease, and progressive disease (PD) is defined as the appearance of endometrial cancer in patients. Continuous therapies will be needed in PR, NR, or PD. Two months of maintenance treatment will be recommended for patients with CR, and participants will be followed up for 2 years.

Outcomes: Primary outcome is the CR rates of the two groups (LNG-IUS alone verse LNG-IUS+ loxenatide) in 16-week. Secondary outcomes include CR rates in 32 weeks, assessment of ovarian functions, improvement of weight, insulin resistance, chronic inflammation condition, and time to achieve CR, and safety and side events during the therapy, and the recurrence rates, pregnancy rates, and live birth rates in two years.

ELIGIBILITY:
Inclusion Criteria:

* BMI (body mass index) ≥28kg/m2
* Consent informed and signed
* Pathologically confirmed as endometrial atypical hyperplasia
* Have a strong desire to reproduce and ask for fertility preservation or those who insist on keeping the uterus despite no reproductive requirements
* Have good compliance and follow-up conditions, and patients are willing to follow up in Obstetrics and Gynecology Hospital of Fudan University in time

Exclusion Criteria:

* Diagnosed as type 2 diabetes
* Diabetic ketoacidosis
* History of acute pancreatitis
* Have a history or family history of medullary thyroid carcinoma; multiple endocrine neoplasia syndrome type 2 (MEN2)
* Combined with severe medical disease or severely impaired liver and kidney function
* Patients with other types of endometrial cancer or other malignant tumors of the reproductive system; patients with breast cancer or other hormone- dependent tumors that cannot be used with progesterone
* Those who require hysterectomy or other methods other than conservative treatment with drugs
* Known or suspected pregnancy
* Currently suffering from pelvic inflammatory disease or diagnosed as pelvic inflammatory disease
* Lower reproductive system infection
* abnormal cervical dysplasia
* Congenital or acquired uterine abnormalities, including fibroids that deform the uterine cavity
* Allergic to any parts of LNG-IUS components
* The uterine cavity is too large (average diameter is over 7cm) or the history of LNG-IUS falling off

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (CR) rates | From date of randomization until the date of CR, assessed up to 16 weeks.
  The 16-week CR rates will be calculated in two groups

SECONDARY OUTCOMES:
32-week complete response (CR) rates | From date of randomization until the date of CR, assessed up to 32 weeks.
  The 32-week complete response rates will be calculated in two groups
weight change | From date of randomization until the date of CR, assessed up to 32weeks.
  weight change in 32-week's intervention, weight will be recorded every month
changing of insulin resistance | From date of randomization until the date of CR, assessed up to 32weeks.
  indicators of insulin resistance will be assessed at baseline and every 12-16 weeks.
change of chronic inflammation status | From date of randomization until the date of CR, assessed up to 32 weeks.
  Change of chronic inflammation indications (tumor necrosis factor (TNF-α), interleukin-1(IL-1), interleukin-6 (IL-6)) in 32 weeks
change of ovarian functions | From date of randomization until 6 months after treatment is over
  AMH (anti-mullerian hormone ) will be assessed at baseline and every 12-16 weeks
Time of pathological complete response (CR) | From date of randomization until the date of CR, assessed up to 2 years
  Time of histologic regression from AEH to proliferative or secretory endometrium
safety and side effects | From date of randomization until the date of CR, assessed up to 2 years
  Adverse events related with Liraglutide and LNG-IUS. Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be recorded, as well as incidence of adverse events.
Relapse rates | up to 2 years after the treatment for each patient
  All enrolled patients will be followed up for 2 years. During the following-up period, if patients recur after complete regression, they will be counted and the number of recurrence will be divided by number of patients followed up, then we can get the relapse rates.Comparison will be performed between two groups.
pregnancy outcomes | up to 2 years after the treatment for each patient
  For patients have a desire for fertility, pregnancies, births and related outcomes will be counted, and the rate of pregnancy will be counted as number of pregnancies/ number of patients trying to fertility in the following period. Comparison will be performed between two groups

CONTACTS AND LOCATIONS:
Overall Officials: XIAOJUN CHEN, PhD, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University
Locations (1):
- Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China